CLINICAL TRIAL: NCT02757794
Title: Long-term Effects of Visual Spatial Working Memory Training Program Performed at Preschool Age in Very Preterm Infants With Visual Spatial Working Memory Deficit. A Randomized Controlled Trial
Acronym: EPIREMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-01; 2016-A00122-49 (Registry Identifier: ID RCB); RCAPHM16_0010 (Other: APHM)
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Children Born Extremely Premature; Disturbance of Visuo-spatial Working Memory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive remediation parents (Active Comparator)
  Interventions: Other: computerized cognitive remediation program
- Remediation standard (Placebo Comparator)
  Interventions: Other: standard remediation

INTERVENTIONS:
Other: computerized cognitive remediation program — a computer program online re-educating the working memory is completed by the parents and the child. The child made a series of interactive exercises accompanied by parents or a practitioner. The exercises are adapted automatically and individually to the performance at each session.
  Arms: Cognitive remediation parents
Other: standard remediation — A speech therapy and / or academic support is realized.
  Arms: Remediation standard

SUMMARY:
Prematurity tends to increase in France in recent years and more children born extremely premature infants survive. If severe impairments have stabilized, the majority of former extremely premature children have neuropsychological disorders and moderate appearance behavior disorder, but with a significant impact both family, school and social persisting into adulthood.

Executive functions (EF), in general, and working memory (MT), in particular, are frequently altered in older children preterm infants compared to controls born at term.

The identification process of loss in certain diseases, as well as improving knowledge of brain functioning, and development with the possibility of neuronal plasticity has led research teams to develop intervention programs focused on process cognitive qualified of "remediation" cognitive (RC). Schematically, the RC is defined as a rehabilitation or altered cognitive functions. MT can be improved by encouraging the operation of the spots mental stimulant. These programs are effective on MT but do not have the expected impact on other FE, language or nonverbal functions (visuospatial). The functional benefit of cognitive remediation remains controversial.

Improving mental functions untrained as nonverbal MT, attention and secondarily learning is possible but still unproven on wide population. Similarly, randomized trials are needed to test this type of cognitive remediation among preschoolers old very premature.

ELIGIBILITY:
Inclusion Criteria:

* Already included in the study EPIPAGE 2, born between 24 and 34 weeks' GA (gestational amenorrhea),
* Children aged 5 to 6 years,
* Children exhibiting a total intellectual quotient >70 from the WPPSI IV (during the 5-year assessment in EPIPAGE 2),
* Children having a visuo-spatial Working Memory impairment defined by a working memory index <85 from the WPPSI IV,
* Children with parents (or legal guardians) authorizing participation in the study and a signed informed consent form,
* Children affiliated with medical insurance.

Exclusion Criteria:

* Children with severe cerebral palsy, based on the Gross Motor Function (GMFCS score >2) and Bimanual Fine Motor Function (BFMF >2) classification system (Elvrum AG 2015, Marois P 2015),
* Children with blindness or amblyopia, defined by a visual acuity <3 (during the 5-year assessment in EPIPAGE 2),
* Children with deafness, as defined by a prescribed hearing aid,
* Children with chromosomal disorder or autistic syndrome,
* Children included in the EPILANG study protocol (an ancillary project to EPIPAGE),
* Children who do not speak French
* Children with parents having no internet connection,
* Triplets.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 166 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Increase of the measuring index visuospatial | 18 months (more or less 2 months) post inclusion
  This index consists of two subtests : block design and object assembly. The average score is 100 with a standard deviation of 15.

SECONDARY OUTCOMES:
Assessment of intellectual functioning | 8 months (more or less 2 months) post inclusion
  award of global IQ
Evaluation of the working memory | 18 months (more or less 2 months) post inclusion
  administering the questionnaire Wechsler Preschool and Primary Scale of Intelligence (WPPSI IV)
evaluation of neuropsychological development of children | 8 months (more or less 2 months) post inclusion
  award of Neuropsychological Assessment test (NEPSY)
Evaluation of language and skills | 8 months (more or less 2 months) post inclusion
  passing the test Communicate, Learn to Read and Write (KEY)
Rating behavior | 8 months (more or less 2 months) post inclusion
  award of Goodman questionnaire (Strengths and Difficulties Questionnaire (SDQ))
Evaluation of parental anxiety | 8 months (more or less 2 months) post inclusion
  award of Spielberger Trait Anxiety Inventory questionnaire
Assessing the quality of a child's life | 8 months (more or less 2 months) post inclusion
  Quality of Life Questionnaire
Evaluation of Education | 8 months (more or less 2 months) post inclusion
  Evaluation of Education is evaluated by the global adaptation school score (GSA) survey

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (18):
- France (18):
  - University Hospital of Lyon, Bron
  - University Hospital of Caen Normandie, Caen
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - Sud Francilien Hospital, Corbeil-Essonnes
  - University Hospital of Grenoble, Grenoble
  - Assistance Publique Hôpitaux de Marseille, Marseille
  - University Hospital of Montpellier, Montpellier
  - Regional University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - University Hospital of Nice, Nice
  - University Hospital of Nîmes, Nîmes
  - AP- HP - Armand Trousseau Hospital, Paris
  - University Hospital of Reims, Reims
  - University Hospital of Rouen, Rouen
  - University Hospital of Saint-Etienne, Saint-Etienne
  - Regional University Hospital of Strasbourg, Strasbourg
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tour, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gire C, Beltran Anzola A, Marret S, Foix L'Helias L, Roze JC, Granier M, Patural H, Lecomte B, Guillois B, Souksi Medioni I, Bednarek Weirauch N, Claris O, Hascoet JM, Kuhn P, Zahed M, Boucekine M, Ancel PY, Arnaud C, Cambonie G, Dorriere Datin V; EPIREMED Study Group. Cognitive Training for Visuospatial Processing in Children Aged 5(1/2) to 6 Years Born Very Preterm With Working Memory Dysfunction: A Randomized Clinical Trial. JAMA Netw Open. 2023 Sep 5;6(9):e2331988. doi: 10.1001/jamanetworkopen.2023.31988. PMID 37676661
- [Derived] Gire C, Beltran Anzola A, Kaminski M, Baumstarck K, Ancel PY, Berbis J; for EPIREMED-Study Group. A randomized EPIREMED protocol study on the long-term visuo spatial effects of very preterm children with a working memory deficit. BMC Pediatr. 2021 Sep 13;21(1):402. doi: 10.1186/s12887-021-02867-x. PMID 34517869